CLINICAL TRIAL: NCT01766518
Title: Open Label, Multicenter, Non-comparative Study to Evaluate the Efficacy and Safety of MY-REPT Capsule in Primary, Liver Transplantation Recipients.
Brief Title: The Study to Evaluate Efficacy and Safety of MY-REPT Capsule in Primary, Liver Transplantation Recipients (MYLT1)
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: m307LTP09D
Record Dates: First submitted 2013-01-10; First posted 2013-01-11 (Estimated); Last update posted 2013-11-07 (Estimated); Status verified 2013-11

CONDITIONS: Evidence of Liver Transplantation
Keywords: liver transplantation; LT; Mycophenolate mofetil; MMF
MeSH Terms: interventions — Mycophenolic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MY-REPT capsule (Experimental): MY-REPT capsule: Mycophenolate mofetil, 250mg/cap, orally
  Interventions: Drug: Mycophenolate mofetil

INTERVENTIONS:
Drug: Mycophenolate mofetil — MY-REPT capsule 500~1500mg/day, per oral, capsules twice a day with Tacrolimus, Corticosteroids, Basiliximab post liver transplantation
  Other Names: MY-REPT capsule

SUMMARY:
Efficacy and safety of MY-REPT capsule in primary, liver transplantation recipients

DETAILED DESCRIPTION:
Open label, Multicenter, Non-comparative Study to evaluate the efficacy and safety of MY-REPT capsule in primary, liver transplantation

ELIGIBILITY:
Inclusion Criteria:

* Patient with primary liver transplantation recipients
* Male and Female aged ≥19 and ≤65
* Patient with ABO blood type correspond with Donor's blood type
* Patient who agreement with written informed consent
* Patient who Women if had childbearing potential must have a negative serum or urine pregnancy test at the screening visit and agreement with contraception

Exclusion Criteria:

* Patient with secondary liver transplantation(LT) recipient or other organ transplantation recipient in past or current
* Patient with multi-organ transplantation recipient
* Patient with dual-graft transplantation recipient
* Patient who used body artificial liver before LT
* Cr level >2.0mg/dL in screening
* WBC <2,000/mm3 or ANC <900/mm3 or PLT <30,000/mm3 in screening
* Patient who experienced severe gastrointestinal disorder so investigator judge the man's participation impossible
* Patient who experienced severe infection (need to treatment)
* Patient or Donor with HIV positive
* Patient who need to treat with immunosuppressant or chemistry therapy
* Patient who had taken immunosuppressant within 30days before LT (except to take Corticosteroids and Tacrolimus due to protocol)

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2009-11; Primary Completion 2014-04 (Estimated); Study Completion 2014-05 (Estimated)

PRIMARY OUTCOMES:
Rate of acute rejection | up to 26weeks
  Rate acute rejection by liver biopsy

SECONDARY OUTCOMES:
Frequency, Time, Severity of acute rejection | up to 26 weeks
Graft loss, Patient survival rate | up to 26weeks
Kidney function test by e-GFR(Glomerular filtration rate) | up to 26weeks
Questionnaire of gastrointestinal symptom assessment | screening visit, closing visit
Questionnaire of gastrointestinal quality of life index | screening visit, closing visit

OTHER OUTCOMES:
Rate of adverse event | up to 26 weeks
Laboratory test | up to 26weeks
Physical exam, pulse rate et. | up to 26weeks

CONTACTS AND LOCATIONS:
Overall Officials: SungGyu Lee, Ph.D, Principal Investigator — Asan Medical Center
Locations (3):
- South Korea (3):
  - Asan medical center, Seoul
  - Samsung Medical Center, Seoul
  - Seoul ST Mary's Hospital, Seoul